CLINICAL TRIAL: NCT00632853
Title: Phase III Comparison of Thoracic Radiotherapy Regimens in Patients With Limited Small Cell Lung Cancer Also Receiving Cisplatin and Etoposide
Brief Title: Radiation Therapy Regimens in Treating Patients With Limited-Stage Small Cell Lung Cancer Receiving Cisplatin and Etoposide
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-30610; CALGB-30610 (Other: Cancer and Leukemia Group B); RTOG 0538 (Other: Radiation Therapy Oncology Group); U10CA031946 (NIH); CDR0000588879 (Registry Identifier: Physician Data Query); NCI-2009-00470 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2008-03-08; First posted 2008-03-11 (Estimated); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Etoposide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A - Standard Radiotherapy + Chemotherapy (Active Comparator): Radiotherapy (every day, Monday-Friday, for a total of 3 weeks) XRT: 45 Gy BID (1.5 Gy/fx) starting on day 1 of Cycle 1 or 2, every day, for 3 weeks
  Chemotherapy (every 21 days for 4 cycles, for a total of 12 weeks):
  * Cisplatin 80 mg/m2 IV on day 1 OR Carboplatin AUC 5 IV day 1, every 21 days
  * Etoposide 100 mg/m2 IV Register/ on days 1, 2, and 3, every 21 days
  Interventions: Radiation: Standard Radiation Dose Therapy; Drug: cisplatin; Drug: etoposide; Drug: carboplatin
- Arm B - High Dose Radiotherapy + Chemotherapy (Experimental): Radiotherapy (every day, Monday-Friday, for a total of 7 weeks) XRT: 70 Gy QD (2.0 Gy/fx), starting on day 1 of Cycle 1 or 2, every day, for 7 weeks
  Chemotherapy (every 21 days for 4 cycles, for a total of 12 weeks):
  * Cisplatin 80 mg/m2 IV on day 1 OR Carboplatin AUC 5 IV day 1, every 21 days
  * Etoposide 100 mg/m2 IV on days 1, 2, and 3, every 21 days
  Interventions: Drug: cisplatin; Drug: etoposide; Radiation: High Radiation Dose Therapy; Drug: carboplatin

INTERVENTIONS:
Radiation: Standard Radiation Dose Therapy — 45 Gy
  Arms: Arm A - Standard Radiotherapy + Chemotherapy
Drug: cisplatin — IV
Drug: etoposide — IV
Radiation: High Radiation Dose Therapy — 70 Gy
  Arms: Arm B - High Dose Radiotherapy + Chemotherapy
Drug: carboplatin — IV

SUMMARY:
Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as etoposide, carboplatin and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known which radiation therapy regimen is more effective when given together with chemotherapy in treating patients with limited-stage small cell lung cancer. This randomized phase III trial is comparing different chest radiation therapy regimens to see how well they work in treating patients with limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a 2-part, multicenter, randomized study. Patients are stratified according to gender, weight loss 6 months prior to study entry (≤ 5% of body weight vs > 5% of body weight), ECOG performance status (0 vs 1 vs 2), radiotherapy technique (intensity-modulated radiotherapy vs 3-dimensional conformal radiotherapy), radiotherapy start time (at first cycle of protocol chemotherapy, after one cycle of prior non-protocol chemotherapy vs at first cycle of protocol chemotherapy, without prior non-protocol chemotherapy vs at second cycle of protocol chemotherapy, without prior non-protocol chemotherapy) and chemotherapy backbone: carboplatin vs cisplatin.

OBJECTIVES:

Primary Objective

To determine whether administering high dose thoracic radiotherapy, 70 Gy (2 Gy once-daily over 7 weeks) or 61.2 Gy (1.8 Gy once-daily for 16 days followed by 1.8 Gy twice-daily for 9 days), will improve median and 2-year survival compared with 45 Gy (1.5 Gy twice-daily over 3 weeks) in patients with limited stage small cell lung cancer.

Secondary Objectives

1. To compare treatment related toxic effects of thoracic radiotherapy regimens in patients with limited stage small cell lung cancer
2. To compare response rates, failure-free survival and toxicity of thoracic radiotherapy regimens in patients with limited stage small cell lung cancer
3. To compare rates of local relapse, distant metastases and brain metastases with these regimens
4. To compare patients' quality of life between these treatment regimens in terms of their physical symptoms, physical functioning and psychological state
5. To describe the patterns of use of thoracic intensity modulated radiation therapy (IMRT) in patients with limited stage small cell lung cancer
6. To examine blood-based biomarkers of response and resistance to cisplatin (or carboplatin) and etoposide
7. To evaluate the correspondence between increases in plasma ProGRP concentrations and disease progression/recurrence
8. To evaluate the potential for plasma ProGRP concentrations at baseline, after each cycle of chemotherapy and at first evaluation following completion of chemotherapy to predict PFS and OS
9. To evaluate the correspondence between longitudinal decreases in plasma ProGRP concentrations and clinical response

Part 1: Patients are randomized to 1 of 3 treatment arms.

Arm I: Patients undergo standard-dose (45 Gy given in 30 treatments) thoracic radiotherapy twice daily, 5 days a week, for 3 weeks. Patients also receive cisplatin IV on day 1 or carboplatin IV and etoposide IV on days 1, 2, and 3.

Arm II: Patients undergo higher-dose (70 Gy given in 35 treatments) thoracic radiotherapy once daily, 5 days a week, for 7 weeks. Patients also receive cisplatin or carboplatin and etoposide as in arm I.

Arm III: (discontinued as of 03/10/13) Patients undergo mid-dose (61.2 Gy given in 34 treatments) thoracic radiotherapy once daily, 5 days a week, during the initial 16 days (approximately 3 weeks) of treatment and then twice daily, 5 days a week, for the final 9 days (approximately 2 weeks) of treatment. Patients also receive cisplatin and etoposide.

In all arms, treatment with cisplatin and etoposide repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Part 2: An interim analysis was conducted after accrual of 30 patients per arm and one experimental arm based upon a comparison of treatment-related toxicity was selected. The most toxic experimental arm was discontinued, and the trial continues comparing standard therapy (arm I) to the selected experimental regimen (arm II) as described in part 1. Please see the Arms section for more information regarding Part 2.

Prophylactic cranial irradiotherapy (PCI): Within 3-6 weeks after completion of chemotherapy, PCI should be offered to all patients with a complete tumor response (CR) or near complete response (nCR) with only residual chest abnormalities of indeterminate nature following completion of combined modality therapy.

After completion of study treatment, patients are followed up at least every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years or until disease progression. At disease progression, patients are followed up every 6 months.

ELIGIBILITY:
1. Documentation of Disease

   1. Histologically or cytologically documented small cell lung cancer (SCLC)
   2. Limited-stage disease patients with disease restricted to one hemithorax with regional lymph node metastases, including ipsilateral hilar, ipsilateral and contralateral mediastinal, and ipsilateral supraclavicular lymph nodes

      * Patients with disease involvement of the contralateral hilar or supraclavicular lymph nodes are not eligible
      * Patients with pleural effusions that are visible on plain chest radiographs, whether cytologically positive or not are not eligible unless they have a negative thoracentesis
      * Patients with cytologically positive pleural or pericardial fluid, regardless of the appearance on plain x-ray are not eligible
2. Measurable disease - Patients must have measurable disease, which includes lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 2 cm with conventional techniques OR ≥ 1 cm by spiral CT scan
3. Prior Treatment

   1. Patients may have received one and only one cycle of chemotherapy prior to enrolling on CALGB 30610, which must have included carboplatin or cisplatin and etoposide.
   2. If a patient has had one cycle of cisplatin or carboplatin/etoposide prior to registration, the patient must have had all of it prior to registration tests as outlined in the protocol and prior to starting their first cycle of chemotherapy.
   3. Additionally, these patients also must have met all of the eligibility criteria in the protocol prior to receiving the first cycle of chemotherapy.
   4. Registration to CALGB 30610 must take place within 14-21 days after the start of the non-protocol therapy.
   5. Failing to do all of the above will make the patient NOT eligible for CALGB 30610.
   6. No prior radiotherapy or chemotherapy (except for the chemotherapy described in the bullet above) for SCLC
   7. No prior mediastinal or thoracic radiotherapy
   8. Patients with complete surgical resection of disease are not eligible
4. Age Requirement ≥ 18 years of age
5. ECOG Performance Status 0-2
6. Non-pregnant and non-nursing - No patients that are known to be pregnant or nursing
7. Required Initial Laboratory Values

   1. Granulocytes ≥ 1,500/µl
   2. Platelet count ≥ 100,000/µl
   3. Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
   4. AST (SGOT) ≤ 2.0 times ULN
   5. Serum creatinine ≤ 1.5 times ULN OR Calculated creatinine clearance ≥ 70 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2022-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Bogart, MD, Study Chair — State University of New York - Upstate Medical University
Locations (934):
- United States (930):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - The Kirklin Clinic at Acton Road, Birmingham, Alabama
  - Providence Hospital, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - 21st Century Oncology-Scottsdale, Scottsdale, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group-Rogers, Rogers, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - Kaiser Permanente Dublin, Dublin, California
  - 21st Century Oncology - El Segundo, El Segundo, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mercy UC Davis Cancer Center, Merced, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - University of Colorado, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - 21st Century Oncology - Bradenton, Bradenton, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - 21st Century Oncology - Fort Walton Beach, Fort Walton Beach, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Integrated Community Oncology Network-Southside Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network-Florida Cancer Center Beaches, Jacksonville Beach, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - 21st Century Oncology - Lakewood Ranch Oncology, Lakewood Rch, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - AdventHealth Medical Group Urology at Orlando, Orlando, Florida
  - AdventHealth Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - 21st Century Oncology-Palatka, Palatka, Florida
  - Integrated Community Oncology Network-Flager Cancer Center, Saint Augustine, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Tanner Medical Center/Carrollton, Carrollton, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Low Country Cancer Care Associates PC, Savannah, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Mason District Hospital, Havana, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Robert Veith MD LLC, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Veterans Administration Medical Center-Baltimore, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Richard A Henson Cancer Institute at Ocean Pines, Ocean Pines, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - Unspecified Site, Rockville, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Steward Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - 21st Century Oncology MHP - Clarkston, Clarkston, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - 21st Century Oncology MHP - Farmington, Farmington Hills, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - 21st Century Oncology MHP - Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Fairview Maple Grove Medical Center, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center - 68th Street Place, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Cancer Care Specialists - Reno, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Norris Cotton Cancer Center-Nashua, Nashua, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - The Valley Hospital-Luckow Pavilion, Paramus, New Jersey
  - Neurosurgeons of New Jersey-Ridgewood, Ridgewood, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Veterans Affairs Western New York Health Care System-Buffalo, Buffalo, New York
  - Sands Cancer Center, Canandaigua, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - Rochester General Hospital, Rochester, New York
  - University Radiation Oncology, Rochester, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Syracuse Veterans Administration Medical Center, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - Mountain Radiation Oncology PA, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Transylvania Regional Hospital, Brevard, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Angel Medical Center, Franklin, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Carolina Radiation Medicine's Cancer Treatment Center, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Lake Norman Hematology Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Vidant Oncology-Kenansville, Kenansville, North Carolina
  - Novant Health Oncology Specialists-Kernersville, Kernersville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Mission Hospital McDowell, Marion, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Lake Norman Hematology Oncology Specialists-Mooresville, Mooresville, North Carolina
  - Novant Health Oncology Specialists-Mount Airy, Mount Airy, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Vidant Oncology-Richlands, Richlands, North Carolina
  - Carolina Oncology Associates PA, Salisbury, North Carolina
  - Rowan Regional Medical Center, Salisbury, North Carolina
  - Blue Ridge Regional Hospital, Spruce Pine, North Carolina
  - Novant Health Oncology Specialists-Statesville, Statesville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - NHRMC Radiation Oncology - Supply, Supply, North Carolina
  - Novant Health Oncology Specialists-Davidson County, Thomasville, North Carolina
  - Novant Health Oncology Specialists-Wilkesboro, Wilkesboro, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - NHRMC Radiation Oncology - 16th Street, Wilmington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Winston-Salem Health Care, Winston-Salem, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Salem Regional Medical Center, Salem, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - University Pointe, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Surgical Associates Inc, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Mid-Columbia Medical Center/Celilo Cancer Center, The Dalles, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Crozer Regional Cancer Center at Brinton Lake, Glen Mills, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Holy Redeemer Hospital and Medical Center, Meadowbrook, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Upper Delaware Valley Cancer Center, Milford, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Jameson, New Castle, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Aria Health-Torresdale Campus, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - Crozer-Chester Medical Center, Upland, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Carolina Regional Cancer Center, Myrtle Beach, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Regional Cancer Center at Indian Path Community Hospital, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Blount Memorial Hospital, Maryville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Baptist Hospitals of Southeast Texas Cancer Center, Beaumont, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Wellmont Medical Associates-Bristol, Bristol, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Rabin Medical Center, Petah Tikva, Israel
- Puerto Rico (2):
  - San Juan Community Oncology Group, San Juan
  - San Juan City Hospital, San Juan
- Yonsei University Health System-Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Farris MK, Mix MD, Wang X, Jaszewski B, Foster N, Masters GA, Laurie F, Smith K, Razavian NB, Alden RS, Komaki R, Stinchcombe TE, Bradley JD, Vokes EE, Bogart J. Prognostic Factors in Limited-Stage Small Cell Lung Cancer: A Secondary Analysis of CALGB 30610-RTOG 0538. JAMA Netw Open. 2024 Oct 1;7(10):e2440673. doi: 10.1001/jamanetworkopen.2024.40673. PMID 39446327
- [Derived] Bogart J, Wang X, Masters G, Gao J, Komaki R, Gaspar LE, Heymach J, Bonner J, Kuzma C, Waqar S, Petty W, Stinchcombe TE, Bradley JD, Vokes E. High-Dose Once-Daily Thoracic Radiotherapy in Limited-Stage Small-Cell Lung Cancer: CALGB 30610 (Alliance)/RTOG 0538. J Clin Oncol. 2023 May 1;41(13):2394-2402. doi: 10.1200/JCO.22.01359. Epub 2023 Jan 9. PMID 36623230
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.cancer.gov/about-cancer/treatment/clinical-trials/search/v?id=NCI-2009-00470&q=CALGB-30610

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Radiotherapy (every day, Monday-Friday, for a total of 3 weeks)> XRT: 45 Gy BID (1.5 Gy/fx) starting on day 1 of Cycle 1 or 2, every day, for 3 weeks> Chemotherapy (every 21 days for 4 cycles, for a total of 12 weeks):>
  * Cisplatin 80 mg/m2 IV on day 1 OR Carboplatin AUC 5 IV day 1, every 21 days>
  * Etoposide 100 mg/m2 IV Register/ on days 1, 2, and 3, every 21 days> Standard Radiation Dose Therapy: 45 Gy
- Arm B: Radiotherapy (every day, Monday-Friday, for a total of 7 weeks)> XRT: 70 Gy QD (2.0 Gy/fx), starting on day 1 of Cycle 1 or 2, every day, for 7 weeks> Chemotherapy (every 21 days for 4 cycles, for a total of 12 weeks):>
  * Cisplatin 80 mg/m2 IV on day 1 OR Carboplatin AUC 5 IV day 1, every 21 days>
  * Etoposide 100 mg/m2 IV on days 1, 2, and 3, every 21 days
- Arm C: Radiotherapy (every day, Monday-Friday, for a total of 5 weeks)> XRT: 61.2 Gy Concomitant boost: QD (1.8 Gy/fx), starting on day 1 of Cycle 1 or 2, every day, for 16> days of treatment; then BID (1.8 Gy/fx) for 9 days of treatment Chemotherapy (every 21 days for 4 cycles, for a total of 12 weeks)> Cisplatin 80 mg/m2 IV on day 1, every 21 days> Etoposide 100 mg/m2 IV on days 1, 2, and 3, every 21 days
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C
Started | 313 | 325 | 93
Completed | 313 | 325 | 93
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Radiotherapy (every day, Monday-Friday, for a total of 7 weeks)> XRT: 45 Gy QD (2.0 Gy/fx), starting on day 1 of Cycle 1 or 2, every day, for 7 weeks> Chemotherapy (every 21 days for 4 cycles, for a total of 12 weeks):>
  * Cisplatin 80 mg/m2 IV on day 1 OR Carboplatin AUC 5 IV day 1, every 21 days>
  * Etoposide 100 mg/m2 IV on days 1, 2, and 3, every 21 days
- Arm C: Radiotherapy (every day, Monday-Friday, for a total of 7 weeks)> XRT: 61.2 Gy QD (2.0 Gy/fx), starting on day 1 of Cycle 1 or 2, every day, for 7 weeks> Chemotherapy (every 21 days for 4 cycles, for a total of 12 weeks):>
  * Cisplatin 80 mg/m2 IV on day 1 OR Carboplatin AUC 5 IV day 1, every 21 days>
  * Etoposide 100 mg/m2 IV on days 1, 2, and 3, every 21 days
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Total
Number analyzed (Participants) | 313 | 325 | 93 | 731
Age, Continuous [Mean (Full Range); unit: years] | 63.3 [42 to 81] | 62.4 [37 to 80] | 61.7 [41 to 77] | 62.7 [37 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 170 | 46 | 375
  Male | 154 | 155 | 47 | 356
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 5 | 25
  Not Hispanic or Latino | 292 | 302 | 85 | 679
  Unknown or Not Reported | 10 | 14 | 3 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 1 | 5
  Asian | 4 | 4 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 27 | 27 | 11 | 65
  White | 271 | 281 | 80 | 632
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 9 | 10 | 0 | 19

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Time
Description: Overall survival time is defined as the time between a patient's registration and death or end of survival follow up.
Time Frame: 11.25 years
Population: All registered patients were included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm A: Radiotherapy (every day, Monday-Friday, for a total of 3 weeks) XRT: 45 Gy BID (1.5 Gy/fx) starting on day 1 of Cycle 1 or 2, every day, for 3 weeks> Chemotherapy (every 21 days for 4 cycles, for a total of 12 weeks):> Cisplatin 80 mg/m2 IV on day 1 OR Carboplatin AUC 5 IV day 1, every 21 days> Etoposide 100 mg/m2 IV Register/ on days 1, 2, and 3, every 21 days Standard Radiation Dose Therapy: 45 Gy
- Arm B: Radiotherapy (every day, Monday-Friday, for a total of 7 weeks) XRT: 70 Gy QD (2.0 Gy/fx), starting on day 1 of Cycle 1 or 2, every day, for 7 weeks> Chemotherapy (every 21 days for 4 cycles, for a total of 12 weeks):> Cisplatin 80 mg/m2 IV on day 1 OR Carboplatin AUC 5 IV day 1, every 21 days> Etoposide 100 mg/m2 IV on days 1, 2, and 3, every 21 days
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 313 | 325 | 93
Months | 28.7 [26.2 to 35.5] | 30.5 [24.4 to 39.6] | 32.3 [21.1 to 44.8]
Statistical Analysis 1: Comparison: Arm A vs Arm B vs Arm C; Test type: Superiority; p = 0.8741, Log Rank

2. Secondary Outcome: Complete and Partial Response Rates
Time Frame: 11.25 years
Reporting Status: Not Posted, anticipated posting 2023-08

3. Secondary Outcome: Failure-free >> Survival
Time Frame: Up to 5 years
Reporting Status: Not Posted

4. Secondary Outcome: To Compare Rates of Local Relapse, Distant Metastases and Brain Metastases With These > Regimens.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2023-08

5. Secondary Outcome: To Compare Patients' Quality of Life Between These Treatment Regimens in Terms of Their > Physical Symptoms, Physical Functioning and Psychological State.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2023-08

6. Secondary Outcome: To Describe the Patterns of Use of Thoracic Intensity Modulated Radiation Therapy (IMRT) in Patients With Limited Stage Small Cell Lung Cancer.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2023-08

7. Secondary Outcome: To Examine Blood-based Biomarkers of Response and Resistance to Cisplatin (or Carboplatin) and Etoposide.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2023-08

8. Secondary Outcome: To Evaluate the Correspondence Between Increases in Plasma ProGRP Concentrations and Disease Progression/Recurrence
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2023-08

9. Secondary Outcome: To Evaluate the Potential for Plasma ProGRP Concentrations at Baseline, After Each Cycle of > Chemotherapy and at First Evaluation Following Completion of Chemotherapy to Predict PFS and OS.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2023-08

10. Secondary Outcome: To Evaluate the Correspondence Between Longitudinal Decreases in Plasma ProGRP Concentrations and Clinical Response.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2023-08

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 15 months and mortality was collected over 140 months.
Groups:
- Arm A; Arm B; Arm C: - Etoposide 100 mg/m2 IV on days 1, 2, and 3, every 21 days
Arm/Group | Arm A | Arm B | Arm C
All-Cause Mortality (participants affected / at risk) | 206/313 | 220/325 | 73/93
Serious Adverse Events (participants affected / at risk) | 4/313 | 11/325 | 4/93
Other Adverse Events (participants affected / at risk) | 292/313 | 296/325 | 87/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=313) | Arm B (N=325) | Arm C (N=93)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1)
Death NOS (General disorders) | 0 (0) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 3 (3) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis(unknown ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=313) | Arm B (N=325) | Arm C (N=93)
Blood disorder (Blood and lymphatic system disorders) | 7 (10) | 7 (12) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 41 (51) | 39 (44) | 11 (13)
Hemoglobin decreased (Blood and lymphatic system disorders) | 246 (681) | 247 (660) | 73 (206)
Hemolysis (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 6 (11) | 8 (8) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (5) | 4 (5) | 4 (4)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 4 (8) | 5 (5) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 7 (13) | 8 (10) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (3) | 0 (0) | 0 (0)
Dry eye syndrome (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (3)
Vision blurred (Eye disorders) | 6 (8) | 4 (4) | 1 (2)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 10 (11) | 2 (4)
Colitis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 22 (34) | 29 (50) | 7 (11)
Diarrhea (Gastrointestinal disorders) | 20 (23) | 26 (35) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (6) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 10 (15) | 11 (21) | 5 (7)
Dysphagia (Gastrointestinal disorders) | 161 (317) | 180 (361) | 52 (120)
Esophageal mucositis (clin exam) (Gastrointestinal disorders) | 2 (4) | 4 (5) | 0 (0)
Esophageal mucositis (funct/sympt) (Gastrointestinal disorders) | 2 (2) | 2 (4) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 177 (358) | 164 (323) | 50 (110)
Esophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 18 (23) | 46 (78) | 8 (8)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 4 (6) | 9 (19) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (clin exam) (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Mucositis oral (funct/sympt) (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 187 (392) | 188 (416) | 62 (142)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 92 (150) | 105 (169) | 44 (72)
Chest pain (General disorders) | 10 (14) | 16 (17) | 1 (2)
Chills (General disorders) | 1 (1) | 2 (3) | 0 (0)
Edema limbs (General disorders) | 6 (7) | 8 (16) | 2 (4)
Fatigue (General disorders) | 66 (141) | 76 (168) | 26 (52)
Fever (General disorders) | 10 (10) | 2 (2) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 2 (2) | 0 (0)
Gait abnormal (General disorders) | 2 (2) | 1 (1) | 0 (0)
General symptom (General disorders) | 1 (1) | 1 (13) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 1 (3) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 8 (10) | 17 (22) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (2) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 11 (26) | 14 (22) | 5 (5)
Immune system disorder (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bladder infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchitis(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis(unknown ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Catheter related infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Colitis, infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Encephalitis infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endocarditis infective(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Esophageal infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Esophageal infection(unknown ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eye infection(unknown ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gingival infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection(gr 0/1/2 ANC) (Infections and infestations) | 11 (12) | 12 (14) | 1 (1)
Infectious colitis(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Kidney infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mucosal infection(unknown ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Opportunistic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis externa(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritoneal infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (5) | 2 (2) | 0 (0)
Pneumonia(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia(gr 3/4 ANC) (Infections and infestations) | 4 (4) | 6 (6) | 2 (2)
Pneumonia(unknown ANC) (Infections and infestations) | 1 (1) | 1 (2) | 1 (1)
Sepsis(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sepsis(unknown ANC) (Infections and infestations) | 7 (9) | 2 (2) | 0 (0)
Sinusitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 3 (3) | 4 (6) | 0 (0)
Soft tissue infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upr aerodigstve trct infctn(unknown ANC) (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Urinary tract infection(gr 3/4 ANC) (Infections and infestations) | 3 (3) | 4 (4) | 1 (1)
Urinary tract infection(unknown ANC) (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Wound infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Aortic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 4 (5) | 15 (27) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 1 (1)
Intraoperative renal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 61 (93) | 90 (148) | 24 (42)
Vascular access complication (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 2 (2)
Activated partial throm time prolonged (Investigations) | 2 (2) | 3 (3) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 6 (12) | 1 (1)
Alkaline phosphatase increased (Investigations) | 4 (6) | 6 (11) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 7 (12) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 2 (2)
CD4 lymphocytes decreased (Investigations) | 3 (6) | 8 (11) | 1 (1)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cardiac troponin T increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 84 (155) | 91 (168) | 20 (37)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Laboratory test abnormal (Investigations) | 4 (6) | 3 (6) | 1 (2)
Leukocyte count decreased (Investigations) | 219 (480) | 236 (559) | 73 (174)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 38 (68) | 52 (109) | 21 (34)
Neutrophil count decreased (Investigations) | 213 (411) | 240 (530) | 71 (168)
Platelet count decreased (Investigations) | 63 (96) | 76 (127) | 21 (38)
Serum cholesterol increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 2 (2) | 0 (0)
Weight loss (Investigations) | 120 (236) | 119 (227) | 41 (86)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 27 (43) | 30 (44) | 15 (17)
Blood glucose increased (Metabolism and nutrition disorders) | 20 (30) | 28 (58) | 7 (15)
Blood uric acid increased (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 105 (158) | 108 (178) | 34 (59)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 1 (4)
Serum albumin decreased (Metabolism and nutrition disorders) | 13 (14) | 14 (28) | 5 (6)
Serum calcium decreased (Metabolism and nutrition disorders) | 5 (6) | 17 (25) | 4 (4)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 21 (32) | 28 (52) | 9 (19)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 4 (5) | 7 (8) | 4 (4)
Serum potassium decreased (Metabolism and nutrition disorders) | 27 (31) | 44 (60) | 15 (20)
Serum potassium increased (Metabolism and nutrition disorders) | 4 (4) | 6 (9) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 34 (45) | 40 (66) | 10 (15)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (8) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (19) | 11 (18) | 4 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 7 (10) | 3 (5)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 10 (12) | 9 (11) | 3 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (5) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (10) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 13 (20) | 17 (26) | 7 (8)
Dysgeusia (Nervous system disorders) | 4 (6) | 7 (13) | 4 (6)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 12 (15) | 14 (30) | 3 (4)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 3 (4) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 55 (113) | 60 (134) | 20 (36)
Radiculitis brachial (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 10 (11) | 8 (11) | 3 (3)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 3 (5) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 5 (9) | 13 (19) | 6 (6)
Confusion (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 9 (13) | 7 (11) | 2 (2)
Insomnia (Psychiatric disorders) | 12 (18) | 11 (22) | 4 (7)
Bladder hemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (5) | 3 (4) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 6 (10) | 5 (6) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (4)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 35 (64) | 37 (81) | 10 (20)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 137 (293) | 164 (354) | 44 (92)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (8) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 13 (15) | 1 (1)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal mucositis (clin exam) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0)
Pharyngeal mucositis (funct/sympt) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 17 (22) | 12 (24) | 7 (7)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 6 (6) | 0 (0)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tracheal mucositis (clin exam) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 24 (54) | 31 (68) | 6 (14)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (6) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (5) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (3) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (8) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (2) | 2 (2) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 3 (6) | 0 (0)
Hypertension (Vascular disorders) | 13 (29) | 17 (32) | 2 (2)
Hypotension (Vascular disorders) | 10 (12) | 14 (20) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 13 (19) | 6 (9) | 7 (8)
Vascular disorder (Vascular disorders) | 2 (2) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT00632853/Prot_SAP_000.pdf